CLINICAL TRIAL: NCT06241664
Title: Prospective Clinical Trial to Demonstrate the Efficacy and Safety of the AEYE-DS Software Device for Automated Diabetic Retinopathy Detection From Digital Fundoscopic Images Obtained With Multiple Fundoscopy Camera Devices
Brief Title: Efficacy and Safety of AEYE Diagnostic Screening (AEYE-DS) Software Device for Detection of Diabetic Retinopathy From Digital Funduscopic Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AEYE Health Inc (Industry)
Collaborators: A. Stein Regulatory Affairs Consulting Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AEYE-DS-003
Record Dates: First submitted 2024-01-21; First posted 2024-02-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Retinopathy, DR; Diabetic Mellitus
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AEYE-DS Software Device (Experimental): Eligible participants will undergo the following procedures: photographic imaging of each eye using various fundoscopy camera devices. Images obtained will be sent to the AEYE-DS software for analysis. Additional photographic and Optical Coherence Tomography (OCT) images will be obtained using a second fundoscopy/OCT camera device. Images obtained will be sent to a professional reading center for analysis. All study subjects will have their pupils dilated using dilation drops.
  Interventions: Device: AEYE-DS Software

INTERVENTIONS:
Device: AEYE-DS Software — An Artificial Intelligence (AI) software device to be used as a diagnostic tool to assist healthcare providers in screening for diabetic retinopathy (DR) using digital funduscopic images. The device automatically detects more than mild diabetic retinopathy (mtmDR) in adults diagnosed with diabetes who have not been previously diagnosed with DR.

SUMMARY:
The goal of this clinical trial is to learn about the performance of the AEYE-DS Software Device to automatically detect more than mild Diabetic Retinopathy (mtmDR) in adult participants diagnosed with Diabetic Mellitus (DM) using fundoscopic images of the eyes. The main question it aims to answer is if the software is effective in diagnosing more than mild Diabetic Retinopathy (mtmDR) in patients with known diabetes using digital funduscopic images, acquired from each of the participating fundoscopy devices and based on one macula centered image per eye.

Participants:

* will have an eye exam in which photographic images of each eye will be taken by a novice operator, using four different FDA approved/registered fundoscopy cameras. These images will be sent to and analyzed by the AEYE-DS software device.
* will have additional eye imaging taken using a different FDA approved desktop camera system by a professional ophthalmic photographer. These images will be sent to an independent reading center for analysis.
* will have dilation drops put in their eyes (either during or after the imaging with the fundoscopy cameras), wait about 30 minutes for the pupils to dilate and continue the eye imaging exams.

The outcome results with the AEYE-DS Software will be compared to the analysis of the eye images processed by the reading center to see if the investigational software device was accurate in its diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Age≥22
* Documented diagnosis of diabetes mellitus, meeting the criteria established by the American Diabetes Association (ADA) and World Health Organization (WHO):

  1. Elevated Hemoglobin A1c (HbA1c) ≥ 6.5% (48mmol/mol), based on repeated assessments, performed in a laboratory using a method that is National Glycohemoglobin Standardization Program (NGSP) certified and standardized to the Diabetes Control and Complications Trial (DCCT) assay OR
  2. Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L), based on repeated assessments, where 'fasting' is defined as no caloric intake for at least 8 hours OR
  3. Oral Glucose Tolerance Test (OGTT) with two hour plasma glucose (2-hr PG) ≥200 mg/dl (11.1 mmol/L), using the equivalent of an oral 75 g anhydrous glucose dose dissolved in water OR
  4. Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dl (11.1 mmol/L)
* Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

* Uncorrectable vision loss (e.g., with the use of eyeglasses), blurred vision, or floaters.
* Diagnosed with macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion.
* Previously diagnosed with Diabetic Retinopathy.
* History of laser treatment of the retina or injections into either eye, or any history of retinal surgery.
* Currently participating in another investigational eye study and actively receiving investigational product for DR or Diabetic Macular Edema (DME).
* Subject has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation).
* Subject is contraindicated for imaging by fundus imaging systems used in the study:

  1. Subject is hypersensitive to light
  2. Subject recently underwent photodynamic therapy (PDT)
  3. Subject is taking medication that causes photosensitivity
  4. Subject has a history of angle-closure glaucoma or narrow anterior chamber angles
* Subject is pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 1 year
  To assess the sensitivity and specificity of the AEYE-DS software device for the detection of more than mild diabetic retinopathy (mtmDR) on digital funduscopic images, acquired from each of the participating fundoscopy devices and based on one macula centered image per eye, in subjects with known diabetes undergoing screening for diabetic retinopathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Network, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No